CLINICAL TRIAL: NCT03327103
Title: Decision Navigation for Advanced Prostate Cancer Treatment Options Using mHealth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: Johns Hopkins University (Other); Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Randy A. Jones, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19402
Record Dates: First submitted 2017-10-26; First posted 2017-10-31 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Decision Support Techniques
Keywords: decision making; advanced prostate cancer; decision aid; minorities; mHealth; community patient navigator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (No Intervention): Receive standard care
- Decision Intervention (Experimental): Receives decision aid intervention that encompasses balance sheets, navigation, audio files, and interaction -- Cancer Health Aid to Manage Preferences and Improve Outcomes through Navigation (CHAMPION)
  Interventions: Behavioral: CHAMPION

INTERVENTIONS:
Behavioral: CHAMPION — An interactive mHealth decision aid that includes immediate and over time quality of life (QL) graphical summaries for advanced prostate cancer patients to enhance informed, shared decision making and will also be used to assess the CPNs' role in the decision-making process.
  Arms: Decision Intervention

SUMMARY:
Prostate cancer is a commonly diagnosed cancer, and is the second leading cause of cancer deaths among men in the U.S. The subgroup of men with advanced prostate cancer is particularly vulnerable to difficult choices for treatment because of the nature of their disease and having limited options. This study will test the use of an innovative Registered Nurse-Community Patient Navigator team delivered interactive mHealth decision aid for patients with advanced prostate cancer to help facilitate informed shared decisions about anti-cancer treatment that affects their quality of life.

DETAILED DESCRIPTION:
Many patients with advanced prostate cancer along with their decision partners/ proxies (DPP) struggle with complex treatment decisions, such as when to start, change, or stop cancer directed treatment. Despite the utility of decision aids (DAs) to address decisional conflict, little is known about treatment decision-making for advanced cancers. The study's primary aim is to test the effects of a theory- based mHealth DA (CHAMPION) administered by Registered Nurse (RN)-Community Patient Navigator (CPN) teams to advanced prostate cancer patients and decision partners/proxies on the following outcomes: less decisional conflict/uncertainty, higher psychosocial quality of life domain (HRQL-PSY), and less regret at the time of making an anti-cancer treatment decision. The secondary aim is to evaluate the CPN role in delivery of the mHealth DA (CHAMPION) from the patients' and decision partners/proxies' perspective. Preliminary estimates of treatment effects by race to see if the data support a larger effect among African Americans versus Others in the primary and secondary aims will also be explored. This mixed-methods population-based randomized controlled trial will gather data from 158 patient/DPP pairs at three sites: University of Virginia Emily Couric Cancer Center, the Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins University, and Virginia Commonwealth University Massey Cancer Center. The pretest/posttest design will measure a time period that includes three single-event decisions over the course of their cancer-directed treatment; and a qualitative retrospective design will allow exploring the experiences of both patients and their DPPs separately in an interview at the completion of the study. Stratification by race (African-American and Caucasian/Other) and decision point (starting vs. changing vs. stopping anticancer treatment) will be used. There will be two groups: the control (enhanced usual care [EUC]) group and the decision intervention (DI) group. The DI group will receive an interactive 7-component cognitive-behavioral skills mHealth program (DA) with a RN-CPN team, primarily focusing on decision-making during cancer treatment. Self-report measures will be used for all participants in addition to probes for the taped interviews with DI. The primary outcome measures are 1) decisional conflict (uncertainty), 2) decisional regret, 3) HRQL-PSY, and 4) decision-making participation preference. Generalized linear models will be used for data analysis for the quantitative component, and qualitative evaluation of the intervention will be conducted to capture each pair's experience of the CHAMPION intervention. This innovative mHealth DA delivered by a CPN is expected to increase acceptability and the uptake of both the DA and the technology components. This addresses several NIH/NINR innovative questions, through the use of information technology to promote health-related decision-making for providers and patients, examining patient outcomes for improvement in healthcare, as well as to engage and support individuals such as extended family, lay coaches, etc. to augment provider care and recommendations.

ELIGIBILITY:
Inclusion Criteria:

* 1) stages III/ IV prostate cancer 2) life expectancy ≥6 months 3) Karnofsky Performance Status >60 4) willingness of a DPP (patient selected person who provides decisional support) to participate 5) pair ages >18 years 6) ability to understand English

Exclusion Criteria:

* severe psychiatric problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2017-07-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Decision Conflict, Decision Regret, and Prostate Cancer Symptom Scale | 9 months
  demonstrate less decisional conflict/uncertainty, higher QL (HRQL-PSY domain) and less regret at the time of making an anti-cancer treatment decision

SECONDARY OUTCOMES:
semi-structured interview | 9 months
  evaluate community patient navigator role in delivery of decision aid

CONTACTS AND LOCATIONS:
Overall Officials: Randy A Jones, PhD,RN,FAAN, Principal Investigator — University of Virginia
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carhuapoma LR, Thayer WM, Elmore CE, Gildersleeve J, Singh T, Shaukat F, Uveges MK, Gray T, Chu C, Song D, Hollen PJ, Wenzel J, Jones RA. Employing a mobile health decision aid to improve decision-making for patients with advanced prostate cancer and their decision partners/proxies: the CHAMPION randomized controlled trial study design. Trials. 2021 Sep 16;22(1):631. doi: 10.1186/s13063-021-05602-0. PMID 34530868